CLINICAL TRIAL: NCT01890057
Title: The Dose of Sugammadex for Rapid Reversal of Profound Neuromuscular Block in Young and Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2013-0280
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Anesthesia Recovery Period, Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Young adults (Experimental): To find out the the dose of sugammadex for recovery of the TOF ratio to 0.9 within 2 minutes from profound neuromuscular block : Dixon's up-and-down method
  Interventions: Drug: Sugammadex
- Elderly adults (Experimental): To find out the the dose of sugammadex for recovery of the TOF ratio to 0.9 within 2 minutes from profound neuromuscular block : Dixon's up-and-down method
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — The dose of sugammadex

SUMMARY:
To find out the dose of sugammadex for recovery of the TOF ratio to 0.9 within 2 minutes from profound rocuronium-induced neuromuscular block in young and elderly adult patients.

DETAILED DESCRIPTION:
A previous study reported that elderly patients required a longer time to recover from rocuronium induced neuromuscular block compared to younger patients. Therefore, the aim of this study is to find out the dose of sugammadex for rapid recovery from profound neuromuscular block in young and elderly adult patients.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years or ≥70 years ASA class I-II patients who received surgery less than 2 hours.

Exclusion Criteria:

* anticipated difficult intubation
* neuromuscular, hepatic or renal disorders
* drug allergy
* body mass index >30 kg/m2 or body mass index <18 kg/m2
* emergency surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The dose of sugammadex for recovery of the TOF ratio to 0.9 within 2 minutes from profound neuromuscular block | 2 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea